CLINICAL TRIAL: NCT02089230
Title: Phase I/II Trial of MEK Inhibitor MEK162 in Patients With Relapsed and or Refractory Acute Myeloid Leukemia and Patients With Poor Prognosis Acute Myeloid Leukemia Not Suitable for or Unwilling to Receive Standard Therapy
Brief Title: MEK Inhibitor 162 Relapsed and/or Refractory Acute Myeloid Leukemia (AML) and Poor Prognosis, Not Suitable for or Unwilling to Receive Standard Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was terminated due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0116; NCI-2014-01518 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia; AML; Advanced leukemias; Myelodysplastic syndrome; MDS; Acute lymphoblastic leukemia; ALL; Relapsed; Refractory; MEK 162
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Cohort 1 - MEK 162 (Experimental): Phase I Starting Dose of MEK 162: 30 mg by mouth twice a day in a 28 day cycle.
  Interventions: Drug: MEK 162
- Phase I Cohort 2 - MEK 162 (Experimental): Phase I Starting Dose of MEK 162: 45 mg by mouth twice a day in a 28 day cycle.
  Interventions: Drug: MEK 162
- Phase II Cohort 3 - MDK 162 (Experimental): Phase II Starting Dose of MEK 162: 45 mg by mouth twice a day in a 28 day cycle.
  Interventions: Drug: MEK 162

INTERVENTIONS:
Drug: MEK 162 — Phase I Starting Dose of MEK 162: 15 mg by mouth twice a day in a 28 day cycle.
  Phase II Starting Dose of MEK 162: Maximum tolerated dose from Phase I.

SUMMARY:
The goal of Phase 1 of this clinical research study is to find the highest tolerable dose of MEK162 that can be given to patients with advanced leukemia.

This is an investigational study. MEK162 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 57 patients total will take part in both phases of this study . All will be enrolled at MD Anderson.

The goal of Phase 2 of this clinical research study is to learn if MEK162 can help to control AML in older patients with advanced leukemia. The safety of this drug will also be studied.

This is an investigational study. MEK162 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 57 patients total will take part in both phases of this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Phase I:

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 2 groups of 3-6 participants will be enrolled in Phase 1 of the study.

If you are enrolled in Phase 1, the dose of MEK162 you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of MEK162. The second group will receive a higher dose of MEK162 than the group before it, if no intolerable side effects were seen. This is designed to find the highest tolerable dose of MEK 162.

Participants in Phase 2 will then receive the highest tolerated dose that was found in Phase 1.

Study Drug Administration:

You will take MEK162 tablets by mouth 2 times a day (about 12 hours apart) every day with a full cup of water.

There are 4 weeks in each study cycle.

Study Visits:

On Day 1 of Cycle 1:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and blood sugar testing.

On Days 4 and 8 of Cycle 1, blood (about 4 teaspoons) will be drawn for routine tests and blood sugar testing.

Sometime during Days 13-27 of each cycle and again on Day 28 of Cycles 2 and beyond, the study staff will call you and ask about any drugs you may be taking and any side effects you may be having. The calls should last less than 10 minutes each time.

On Day 28 of Cycle 1, you will have a bone marrow aspirate and/or biopsy to check the status of the disease and for biomarker and cytogenetic testing. If bone marrow cannot be collected, blood (about 1-2 teaspoons) will be drawn for these tests.

You will have an EKG and either an ECHO or MUGA scan to check your heart function.

On Day 1 of Cycle 2 and beyond:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and blood sugar testing.
* Urine will be collected for routine tests.
* You will have an eye exam by an eye doctor.
* If you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

On visits when you have blood sugar testing, you should fast for at least 8 hours before the blood draw.

On visits when you have urine collected, you will be given containers to collect your urine over 24 hours if the doctor thinks it is needed.

If it is more convenient to you, you may be able to have some of your blood draws done away from MD Anderson. The study staff will discuss this with you.

Every two or three months during your treatment, you will have an echocardiogram (ECHO) or a multigated acquisition (MUGA) scan to check your heart function.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit.

End-of-Treatment Visit:

After your last dose of study drug:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests
* If the doctor thinks it is needed, you will have a bone marrow aspirate and/or biopsy to check the status of the disease and for biomarker, PD, and/or cytogenetic testing. If you have already had a bone marrow aspirate and/or biopsy recently and your doctor thinks repeating it is not needed, leftover bone marrow will be used for these tests. If bone marrow cannot be collected, blood (about 1-2 teaspoons) will be drawn for these tests.
* You will have an EKG.

Phase II:

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 42 participants will be enrolled in Phase 2 of the study.

Participants in Phase 1 were given a dose of MEK162 based on when they joined the study. Groups of participants were given different dose levels until the highest tolerable dose of MEK162 was found.

If you are enrolled in Phase 2, you will receive MEK162 at the highest dose that was tolerated in Phase 1.

Study Drug Administration:

You will take MEK162 tablets by mouth 2 times a day (about 12 hours apart) every day with a full cup of water.

There are 4 weeks in each study cycle.

Study Visits:

On Day 1 of Cycle 1:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and blood sugar testing.

On Days 4 and 8 of Cycle 1, blood (about 4 teaspoons) will be drawn for routine tests and blood sugar testing.

Sometime during Days 13-27 of each cycle and again on Day 28 of Cycles 2 and beyond, the study staff will call you and ask about any drugs you may be taking and any side effects you may be having. The calls should last less than 10 minutes each time.

On Day 28 of Cycle 1, you will have a bone marrow aspirate and/or biopsy to check the status of the disease and for biomarker and cytogenetic testing. If bone marrow cannot be collected, blood (about 1-2 teaspoons) will be drawn for these tests.

You will have an EKG and either an ECHO or MUGA scan to check your heart function.

On Day 1 of Cycle 2 and beyond:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests and blood sugar testing.
* Urine will be collected for routine tests.
* You will have an eye exam by an eye doctor.
* If you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

On visits when you have blood sugar testing, you should fast for at least 8 hours before the blood draw.

On visits when you have urine collected, you will be given containers to collect your urine over 24 hours if the doctor thinks it is needed.

If it is more convenient to you, you may be able to have some of your blood draws done away from MD Anderson. The study staff will discuss this with you.

Every two or three months during your treatment, you will have an echocardiogram (ECHO) or a multigated acquisition (MUGA) scan to check your heart function.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit.

End-of-Treatment Visit:

After your last dose of study drug:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests
* If the doctor thinks it is needed, you will have a bone marrow aspirate and/or biopsy to check the status of the disease and for biomarker, PD, and/or cytogenetic testing. If you have already had a bone marrow aspirate and/or biopsy recently and your doctor thinks repeating it is not needed, leftover bone marrow will be used for these tests. If bone marrow cannot be collected, blood (about 1-2 teaspoons) will be drawn for these tests.
* You will have an EKG.

ELIGIBILITY:
Inclusion Criteria:

1. PHASE I -- a. Primary or secondary AML according to World Health Organization (WHO) classification, with relapsed or refractory disease or newly diagnosed older subjects (greater than or equal to 65 years of age), not candidates for intensive chemotherapy; b. Subjects with MDS, International Prognostic Scoring System (IPSS) Int-2 or high risk (RAEB-2 only, i.e. greater than or equal to 10% blast) who are resistant or intolerant to standard treatment and are not candidates for transplantation; c. Subjects with ALL, relapsed, refractory or intolerant to standard treatment and for whom no effective treatment options are available.
2. Age greater or equal to 18 years.
3. Patients should be willing and able to give informed consent.
4. Eastern Cooperative Group (ECOG) PS less than or equal to 2.
5. PHASE II -- Patients aged 60 and older with newly diagnosed primary or secondary AML according to WHO classification, without any prior therapy for AML with the exception of (a) emergency Leukapheresis and (b) emergency treatment for hyperleukocytosis with hydroxyurea that is allowed until 24 hours before start of the trial treatment. Note: Prior therapy for preexisting hematological condition e.g. MDS or Myeloproliferative Disorder (MPD), including but not limited to hypomethylating agents is allowed until at least 2 weeks have elapsed from completion of that agent before the first dose of MEK 162.
6. Patients must meet at least one of the following conditions: a. Age greater than or equal to 75 years; b. Age greater or equal to 60 and less than 75 years with at least one of the following poor prognostic factors: i. Secondary AML, as determined by known and documented exposure to chemotherapy or radiation therapy; ii. antecedent history of MDS or myeloproliferative disorder according to WHO criteria for at least 3 months prior to trial entry; iii. unfavorable cytogenetic abnormalities including chromosome 5 and 7 as well as complex; iv. ECOG Performance status 2. (Phase II ONLY)
7. Patients are willing and able to give informed consent. (Phase II only)
8. Only patients with mutated RAS (KRAS and NRAS) mutations are eligible to participate. (Phase II only)
9. Adequate cardiac function defined as: --left ventricular ejection fraction (LVEF) greater than or equal to 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram; -- QTcF interval less than or equal to 480 ms. (Phase II only)

Exclusion Criteria:

1. PHASE I and II -- Administration of any antineoplastic therapy within at least 4 weeks (cytotoxic chemotherapy) or 2 weeks (biological and targeted therapy; hypomethylating agents are considered to be biological therapy) of that therapy of the first MEK 162/MEK 162 dose; except the use of hydroxyurea which can be administered up to 5 g/day up to 24 hours before the initiation of the study drug.
2. Patients should not have received an investigational agent for at least 2 weeks prior to the first study drug dose.
3. Clinical evidence of active Central Nervous System (CNS) leukemia requiring active therapy; prior CNS leukemia well-controlled by ongoing therapy is allowed.
4. Active and uncontrolled infection including but not limited to known infection with HIV, active hepatitis B, or hepatitis C.
5. Major surgery within two weeks prior to trial entry.
6. Liver function tests above the following limits at the screening: total bilirubin > 1.5 x Upper Limit of Normal (ULN) unless related to Gilbert's syndrome or hemolysis, AST and/or ALT > 2.5 X ULN, or for subjects with liver involvement Aspartate Aminotransferase (AST) and/or Alanine transaminase (ALT) > 5 x ULN.
7. Serum creatinine > 1.5 x ULN and/or Creatinine Clearance (CrCl) < 30 mL/min at screening (calculation according to Cockcroft & Gault formula).
8. Pregnant or nursing (lactating) women;
9. Female patients of childbearing potential and male patients with partners of childbearing potential who are not willing ot use highly effective methods of contraception throughout the study and for 1 month after study drug discontinuation. Highly effective contraception methods include: **Total abstinence; or **Male or female sterilization; **Combination of any two of the following (a+b or a+c or b+c); a. Use of oral, injected, or implanted hormonal methods of contraception; b. Placement of an intrauterine device (IUD) or intrauterine system (IUS); c. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
10. Female patients with reproductive potential who do not have a negative blood or urine pregnancy test at screening;
11. History of significant difficulty swallowing, malabsorption or other chronic gastro-intestinal disease or conditions that may hamper compliance and/or absorption of the tested product.
12. Has significant cardiac conduction abnormalities and/ or pacemaker or any of the following criteria: -- History of acute coronary syndromes (including myocardial infarction, unstable angina, Coronary Artery Bypass Grafting (CABG), coronary angioplasty, or stenting) <6 months prior to screening, --Symptomatic chronic heart failure; evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening --Uncontrolled arterial hypertension, defined as BP > 140/100 mmHg (average of 3 consecutive readings)
13. History or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO).
14. Any ophthalmopathy visible at screening that would be considered a risk factor for CSR or RVO by the ophthalmologist (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus, history of hyperviscosity or hypercoagulability syndromes).
15. Subjects with active other tumors, except early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN).
16. Patients who have neuromuscular disorders that are associated with elevated Creatinine Kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
17. Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. NB: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on MEK162 treatment.
18. Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 9/2014 to 9/2017
Period: Overall Study
Arm/Group | Phase I Cohort 1 - MEK 162 | Phase I Cohort 2 - MEK 162 | Phase II Cohort 3 - MDK 162
Started | 3 | 4 | 12
Completed | 3 | 4 | 6
Not Completed | 0 | 0 | 6
Not completed — Death | 0 | 0 | 2
Not completed — Seeking Alternative Therapy | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Cohort 1 - MEK 162 | Phase I Cohort 2 - MEK 162 | Phase II Cohort 3 - MDK 162 | Total
Number analyzed (Participants) | 3 | 4 | 12 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 7 | 11
  >=65 years | 1 | 2 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 57 [33 to 74] | 63 [31 to 77] | 64.5 [33 to 85] | 64 [31 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 1 | 2 | 9 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 4 | 8 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of MEK 162 in Participants With Advanced Leukemias
Description: Maximum tolerated dose is the highest dose level in which <2 patients of 6 develop dose limiting toxicity (DLT).
Time Frame: 28 days
Population: Maximum Tolerated Dose (MTD) was not done for the Phase II portion of the study, therefore 0 participants in the Phase II portion of the study were analyzed.
Measure: Number; unit: Milligrams (mg)
Arm/Group | Phase I Cohort 1 - MEK 162 | Phase I Cohort 2 - MEK 162 | Phase II Cohort 3 - MDK 162
Number analyzed (Participants) | 3 | 4 | 0
Milligrams (mg) | NA — The MTD was not determined until cohort 2 of this study | 45 |

2. Secondary Outcome: Number of Participants With a Response
Description: Response is Complete Remission (CR) or CR with incomplete blood count recovery (CRi) according to International Working Group (IWG) consensus criteria for treatment response in Acute Myeloid Leukemia (AML) (modified): Morphological Complete Remission (CR): Normalization of the peripheral blood absolute neutrophil count > 1.0x109/L, platelets > than 100x109/L no residual evidence of extramedullary disease and bone marrow aspirate with ≤ 5% blasts, no blasts with Auer rods (AML only); and Morphological Complete Remission with incomplete blood count recovery (CRi): Same as CR but without normalization of the peripheral blood absolute neutrophil and platelet count.
Time Frame: Assessed after one 28-day cycle of treatment
Population: Six participants in Phase II Cohort 3 were not evlauable for response.
Measure: Number; unit: participants
Arm/Group | Phase I Cohort 1 - MEK 162 | Phase I Cohort 2 - MEK 162 | Phase II Cohort 3 - MDK 162
Number analyzed (Participants) | 3 | 4 | 6
participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Phase I Cohort 1 - MEK 162 | Phase I Cohort 2 - MEK 162 | Phase II Cohort 3 - MDK 162
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/4 | 8/12
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 10/12
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cohort 1 - MEK 162 (N=3) | Phase I Cohort 2 - MEK 162 (N=4) | Phase II Cohort 3 - MDK 162 (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Progressive Disease (General disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (5)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (5) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Lung Infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Neoplasms Benign, Malignant and Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cohort 1 - MEK 162 (N=3) | Phase I Cohort 2 - MEK 162 (N=4) | Phase II Cohort 3 - MDK 162 (N=12)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alkaline Phosphatase Increase (Investigations) | 2 (2) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Blood Bilirubin Increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Eye Disorders (Eye disorders) | 2 (4) | 2 (2) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT02089230/Prot_SAP_ICF_000.pdf